CLINICAL TRIAL: NCT05125575
Title: Open, Comparative, Randomized, Crossover, Single Dose Bioequivalence Study of Metformin 1000 mg Prolonged Release Tablets (JSC Farmak, Ukraine) vs Glucophage® XR 1000 mg Prolonged Release Tablets in Healthy Subjects Under Fed Conditions.
Brief Title: Fed Bioequivalence Study of 2 Metformin 1000 mg Prolonged Release Tablets in 28 Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joint Stock Company "Farmak" (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FK/MTF/FD
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Pharmacokinetics
Keywords: bioequivalence; pharmacokinetics; generic drugs; Metformin 1000 mg Prolonged Release Tablets; Metformin; Prolonged Release Tablets
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Test Product Metformin 1000 mg Prolonged Release Tablets (JSC Farmak, Ukraine)
  Interventions: Drug: Metformin 1000 mg Prolonged Release Tablets (JSC Farmak, Ukraine)
- Treatment B (Active Comparator): Reference Product Glucophage® XR 1000 mg Prolonged Release Tablets (Merck Serono Ltd, UK)
  Interventions: Drug: Glucophage® XR 1000 mg Prolonged Release Tablets

INTERVENTIONS:
Drug: Metformin 1000 mg Prolonged Release Tablets (JSC Farmak, Ukraine) — One tablet of the Test (T) product was administered orally with 240 mL of water.
  Other Names: Diaformin ® SR
  Arms: Treatment A
Drug: Glucophage® XR 1000 mg Prolonged Release Tablets — One tablet of the Reference (R) product was administered orally with 240 mL of water.
  Other Names: Glucophage® XR
  Arms: Treatment B

SUMMARY:
This study was designed to compare the bioavailability of the Test Product Metformin 1000 mg Prolonged Release Tablets (JSC Farmak, Ukraine) and Reference Product Glucophage® XR 1000 mg Prolonged Release Tablets (Merck Serono Ltd, UK) in healthy male and female volunteers under fed conditions.

DETAILED DESCRIPTION:
An Open, Comparative, Randomized, Crossover Clinical Trial to Evaluate the Bioequivalence of Single Doses of Test Product Metformin 1000 mg Prolonged Release Tablets (JSC Farmak, Ukraine) and Reference Product Glucophage® XR 1000 mg Prolonged Release Tablets (Merck Serono Ltd, UK) in Healthy, Adult Male and Female Subjects Under Fed Conditions.

During each period 21 blood samples were taken: prior to dosing (-1.0) and 1.0, 2.0, 3.0, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5, 7.0, 7.5, 8.0, 8.5, 9.0, 10.0, 12.0, 16.0, 24.0, 32.0 and 36.0 hours after IMP administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and non-pregnant and no breast-feeding females (must have a negative pregnancy test result prior to dosing), Caucasian race.
* Non-smoker or past-smoker (who has stopped smoking at least 6 months before the first dosing).
* Body Mass Index (BMI) 18.5 to 30.0 kg/m2, inclusive and body weight between 50 kg and 100 kg(on the day of screening).
* Subject was available for the whole study and had provided his/her written informed consent.
* Subjects in good health, as determined by screening medical history, physical examination, vital signs assessments (pulse rate, systolic and diastolic blood pressure, and body temperature) and 12-lead ECG (electrocardiogram). Minor deviations outside the reference ranges were acceptable, if deemed not clinically significant by the Investigator.
* Subjects in good health, as determined by screening clinical laboratory evaluations. Minor deviations outside the reference ranges were acceptable, if deemed not clinically significant by the Investigator.
* Acceptance of use of contraceptive measures during the whole study by both female and male subjects.

Exclusion Criteria:

* Known cardiovascular disease, history of hypotension.
* Factors in the subject's history that might predispose to ketoacidosis (including pancreatic insulin deficiency, history of pancreatitis, caloric restriction disorders, restricted food intake, alcohol abuse)
* Gastrointestinal, renal or hepatic diseases and/or pathological findings present or in history, which might interfere with the drug pharmacokinetics.
* Previous liver disease with elevations in serum transaminases.
* Acute or chronic diseases and/or clinical finding which might interfere with the aims of the study or with the drug's safety, tolerability, bioavailability and/or pharmacokinetics of the Investigational Medicinal Product (IMP).
* History of kidney disease and with impaired renal function.
* History of severe allergy or allergic reactions to the study IMP, its excipients or related drugs.
* Clinically significant illness within 28 days before the first dosing, including major surgery.
* Any significant clinical abnormality including Hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV), and / or (human immunodeficiency virus) HIV. (On screening)
* Positive screening urine drugs abuse test or/and alcohol breath test or urine cotinine test, and positive pregnancy test on screening.
* Serious mental disease and/or inability to cooperate with clinical team.
* Sitting blood pressure after a minimum of 5 minutes of rest is out of the range of 100-140 mmHg for systolic blood pressure (BP) and/or 60-100 mmHg for diastolic BP and/or heart rate out of the range of 50-100 bpm during the screening procedure.
* Body ear temperature was out of the range of 35.7-37.6°C at screening.
* Orthostatic hypotension during the screening procedure.
* Drug, alcohol (of ≥ 40 g per day pure ethanol), solvents or caffeine abuse.
* Use of organ-toxic drugs or systemic drugs known to substantially alter liver metabolism within 90 days before the first dosing.
* Use of any prescription medication for a period of 28 days before the first dosing.
* Any systemic over-the-counter (OTC) drug treatment and/or vitamins and/or herbal treatment/or food supplements within 14 days before the first dosing.
* Getting a tattoo, body piercing or any cosmetic treatment involving skin piercing within 90 days before the screening unless evaluated by Investigator as non-significant for inclusion in the study.
* Donation or loss of at least 500 mL of blood within 90 days or donation of plasma or platelets within 14 days before the first dosing.
* Anaemia, haemoglobin below 120 g/L for women and 130 g/L for men at screening.
* Less than 30 days between exit procedure in previous study and the first dosing in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2019-01-19 (Actual); Study Completion 2019-01-19 (Actual)

PRIMARY OUTCOMES:
Cmax | up to 36 hours post-administration
  maximum plasma concentration observed (Cmax)
AUC0-t | up to 36 hours post-administration
  Area under the plasma concentration versus time curve calculated by the trapezoidal rule from sampling time zero to sampling time of the last measurable plasma concentration (AUC0-t)

SECONDARY OUTCOMES:
AUC0-∞ | up to 36 hours post-administration
  Area under the plasma concentration versus time curve from time zero to infinity (AUC0-∞)
tmax | up to 36 hours post-administration
  The time of the maximum plasma concentration (tmax).
λz | up to 36 hours post-administration
  Apparent first-order elimination (λz)
t1/2 | up to 36 hours post-administration
  the elimination or terminal half-life (t1/2)
AUCres | up to 36 hours post-administration
  Residual area AUCres = 100 (AUC0-∞ - AUC0-t) / AUC0-∞ [%]

CONTACTS AND LOCATIONS:
Overall Officials: Vlad Udovytskyi, Study Chair — Joint Stock Company "Farmak"
Locations (1):
- QUINTA-ANALYTICA s.r.o., Prague, Czechia

IPD SHARING:
Plan to Share IPD: No